CLINICAL TRIAL: NCT06206733
Title: A Phase III Study Evaluating the Efficacy and Safety of ASKB589 Combined With CAPOX and PD-1 Inhibitor as First-Line Treatment in Claudin18.2 Positive Patients With Unresectable Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: ASKB589 in Combination With CAPOX and PD-1 Inhibitor in Patients With Advanced or Metastatic GC/GEJ Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AskGene Pharma, Inc. (Industry)
Collaborators: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASK-LC-B589-III-1
Record Dates: First submitted 2023-12-12; First posted 2024-01-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Gastric Adenocarcinoma
Keywords: CLDN 18.2; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; ASKB589
MeSH Terms: interventions — Oxaliplatin; Capecitabine; tislelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Treatment with intravenous infusion of ASKB589 on day 1 of each cycle. The infusion duration should be at least 3 hours, and can be shortened or extended in subsequent cycles as appropriate according to the patient's tolerability. Interruption or slow down of intravenous infusion is allowed to manage toxicity. Dosing is continued every cycle until participants meet the criteria of treatment discontinuation.
  Interventions: Drug: ASKB589; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Tislelizumab
- Group B (Placebo Comparator): Treatment with intravenous infusion of placebo on day 1 of each cycle. The infusion duration should be at least 3 hours, and can be shortened or extended in subsequent cycles as appropriate according to the patient's tolerability. Interruption or slow down of intravenous infusion is allowed to manage toxicity. Dosing is continued every cycle until participants meet the criteria for treatment discontinuation.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Tislelizumab; Drug: Placebo

INTERVENTIONS:
Drug: ASKB589 — ASKB589 will be administered as a minimum 3-hour IV infusion
  Arms: Group A
Drug: Oxaliplatin — Oxaliplatin will be administered as a minimum 2-hour IV infusion
Drug: Capecitabine — Capecitabine will be administered orally twice daily (bid).
Drug: Tislelizumab — Tislelizumab will be administered every 3 weeks Intravenous infusion on day 1 of each cycle.
Drug: Placebo — Placebo will be administered as a minimum 3-hour IV infusion
  Arms: Group B

SUMMARY:
This study is a multicenter, randomized, double-blind, standard-of-care controlled phase III clinical study conducted in China. The purpose of this study is to evaluate the efficacy of ASKB589 plus CAPOX and PD-1 inhibitor compared with placebo plus CAPOX and PD-1 inhibitor (as first-line treatment) as measured by Progression Free Survival (PFS).

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, standard-of-care controlled phase III clinical study conducted in China. The purpose of this study is to evaluate the efficacy of ASKB589 plus CAPOX and PD-1 inhibitor compared with placebo plus CAPOX and PD-1 inhibitor (as first-line treatment) as measured by Progression Free Survival (PFS).

This study will also evaluate efficacy, physical function, safety, and tolerability of ASKB589, as well as its effects on quality of life. Pharmacokinetics (PK) of ASKB589 and the immunogenicity profile of ASKB589 will be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of gastric and gastroesophageal junction
2. Advanced recurrent or metastatic disease confirmed by imaging within 28 days prior to randomization
3. Suitable for chemotherapy combined with PD-1 inhibitor
4. Not suitable for anti-HER2 therapy
5. Have at least one measurable lesion according to RECIST1.1 assessed by site investigator within 28 days prior to randomization
6. CLDN 18.2 positive

Exclusion Criteria:

1. Patients with active central nervous system (CNS) metastases or suspected carcinomatous meningitis
2. Participants have significant gastric bleeding
3. The presence of clinically uncontrollable third interspace fluid
4. Received anti-CLDN18.2 antibody at any time in the past
5. Suspected complete or partial obstruction of gastroesophageal access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Until disease progression or withdrawal from the study (generally up to 24 months)
  PFS is defined as the time from the date of randomization until the date of radiological progressive disease (per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 by Independent Review Committee (IRC)) or death from any cause, whichever is earliest.

SECONDARY OUTCOMES:
Overall Survival (OS) | Until death or withdrawal from the study
  OS is defined as the time from the date of randomization until the date of death from any cause.

OTHER OUTCOMES:
Objective Response Rate (ORR) | Until disease progression or withdrawal from the study (generally up to 24 months)
  ORR is defined as the proportion of participants who have a best overall response of Complete Response (CR) or Partial Response (PR) as assessed by Independent Review Committee (IRC) per RECIST 1.1.
Duration Of Response (DOR) | Until disease progression or withdrawal from the study (generally up to 24 months)
  DOR, defined as the time from the date of the first response (CR/PR) until the date of progressive disease as assessed by IRC per RECIST 1.1 or date of death from any cause, whichever is earliest.
Safety and tolerability assessed by adverse events (AEs) | Until 90 days after the end of treatment
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Number of participants with laboratory assessments abnormalities | Until the end of treatment (generally up to 24 months)
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital signs abnormalities and/or adverse events | Until 90 days after the end of treatment
  Number of participants with potentially clinically significant vital sign values.
Health Related Quality of Life (HRQoL) measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core Questionnaire (EORTC-QLQ-C30) | Until the end of treatment (generally up to 24 months)
  EORTC-QLQ-C30 is a cancer-specific 30-item questionnaire. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change
Health Related Quality of Life (HRQoL) measured by the Global Pain (GP) questionnaire | Until the end of treatment (generally up to 24 months)
  The GP instrument is a single assessment of overall pain where 0 equals no pain and 10 equals extreme pain. Low pain scores are considered a better outcome than a high pain score
Health Related Quality of Life (HRQoL) measured by the EuroQOL Five Dimensions Questionnaire 5L (EQ-5D-5L) questionnaire | Until the end of treatment (generally up to 24 months)
  The EQ-5D-5L is a standardized instrument developed by the EuroQol Group for use as a generic, preference-based measure of health outcomes. The EQ-5D-5L is a 5-item self-reported measure of functioning and wellbeing, which assesses 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension comprises 5 levels (no problems, slight problems, moderate problems, severe problems, extreme problems). A unique EQ-5D-5L health state is defined by combining 1 level from each of the 5 dimensions. This questionnaire also records the respondent's self-rated health status on a vertical graduated (0 = the worst health a participant can imagine to 100 = the best health a participant can imagine) visual analogue scale. Responses to the 5 items will also be converted to a weighted health state index (utility score) based on values derived from general population samples.
Pharmacokinetics (PK) of ASKB589 | up to 6 cycles (21 days for 1 cycle)
  Ctrough will be derived from the PK serum samples collected.
Number of anti-drug antibody (ADA) Positive Participants | up to 6 cycles (21 days for 1 cycle)
  Immunogenicity will be measured by the number of participants that are ADA positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing cancer hospital, Beijing, China